CLINICAL TRIAL: NCT02111096
Title: A Phase 2, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of LY2409021 Compared to Sitagliptin in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study of LY2409021 in Participants With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The overall benefit-risk profile did not support continued development of LY2409021 for type 2 diabetes.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 15286; I1R-MC-GLDJ (Other: Eli Lilly and Company); 2013-004275-12 (EudraCT Number)
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — adomeglivant; Sitagliptin Phosphate; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2409021 (Experimental): 20 milligrams (mg) LY2409021 given orally once daily in the morning for 12 months (52 weeks). Participants remain on stable doses of metformin and sulfonylurea, as prescribed by their personal physician.
  Interventions: Drug: LY2409021; Drug: Metformin; Drug: Sulfonylurea
- Sitagliptin (Active Comparator): 100 mg sitagliptin given orally once daily in the morning for 12 months (52 weeks). Participants remain on stable doses of metformin and sulfonylurea, as prescribed by their personal physician.
  Interventions: Drug: Sitagliptin; Drug: Metformin; Drug: Sulfonylurea
- Placebo (Placebo Comparator): Placebo matching LY2409021 and sitagliptin given orally once daily in the morning for 12 months (52 weeks). Participants remain on stable doses of metformin and sulfonylurea, as prescribed by their personal physician.
  Interventions: Drug: Placebo; Drug: Metformin; Drug: Sulfonylurea

INTERVENTIONS:
Drug: LY2409021 — Administered orally
  Arms: LY2409021
Drug: Sitagliptin — Administered orally
  Arms: Sitagliptin
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Metformin — Administered orally
Drug: Sulfonylurea — Administered orally

SUMMARY:
The intent of this study is to assess the safety of LY2409021 in participants with Type 2 diabetes mellitus taking metformin and sulfonylurea as prescribed by their personal physician. The study treatment is expected to last 12 months (52 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Have been treated with a stable dose of metformin for at least 3 months and have been treated with an optimally effective and stable dose of an sulfonylurea for at least 6 months prior to screening.
* HbA1c value between 7.0% and 10.0%, inclusive.
* Body mass index (BMI) between 20 and 45 kilograms/square meter (kg/m^2), inclusive.

Exclusion Criteria:

* Known type 1 diabetes mellitus.
* More than 1 episode of severe hypoglycemia within 6 months prior to screening.
* Two or more emergency room visits or hospitalizations due to poor glucose control in the 6 months prior to screening.
* Severe gastrointestinal disease that may significantly impact gastric emptying or motility or having undergone gastric bypass or gastric banding surgery.
* Previous history or active diagnosis of pancreatitis.
* Positive hepatitis B surface antigen or hepatitis C antibody.
* Clinical signs or symptoms of liver disease, or hepatic aminotransferases (aminotransferase or alanine aminotransferase) greater than 2.0× upper limit of normal (ULN) or elevated alkaline phosphatase (greater than ULN) unrelated to bone metabolic disease.
* Elevated total bilirubin level (greater than ULN), clinically suspicious signs/symptoms of cirrhosis or history of cirrhosis.
* Current diagnosis, personal history of neuroendocrine tumors, family history of any type of multiple endocrine neoplasia (MEN), or Von Hippel-Lindau.
* Contraindications for magnetic resonance imaging.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (33):
- United States (26):
  - John Muir Health Network - The Osteoporosis Center, Concord, California
  - Valley Endocrine, Fresno, Fresno, California
  - National Research Institute, Los Angeles, California
  - Suncoast Research Group, LLC, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - University of Hawaii, Honolulu, Hawaii
  - East West Medical Institute, Honolulu, Hawaii
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Cedar-Crosse Research Center, Chicago, Illinois
  - Midwest CRC, Crystal Lake, Illinois
  - Iderc, P.L.C., Des Moines, Iowa
  - Cotton O'Neil Clinic, Topeka, Kansas
  - Centex Studies, Inc, Lake Charles, Louisiana
  - Cosmopolitan International Diabetes Center, Columbia, Missouri
  - Mercy Medical Research Institute, Springfield, Missouri
  - Palm Research Center, Las Vegas, Nevada
  - SHS Clinical Research Group, Toms River, New Jersey
  - Office:Alwine,Lk, Downingtown, Pennsylvania
  - University Diabetes and Endocrine Consultants, Chattanooga, Tennessee
  - Dallas Diabetes Endocrine Center, Dallas, Texas
  - Galenos Research, Dallas, Texas
  - San Gabriel Clinical Research, Georgetown, Texas
  - Oakwell Clinical Research, San Antonio, Texas
  - Victorium Clinical Research, San Antonio, Texas
  - Polyclinic, Seattle, Washington
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Puerto Rico (3):
  - PRADNET, Inc. Centro Especializado de Nutricion y Bariatria, Hato Rey
  - American Telemedicine Center, San Juan
  - GCM Medical Group PSC, San Juan
- Taiwan (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changhua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yong Kung City

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Kazda CM, Frias J, Foga I, Cui X, Guzman CB, Garhyan P, Heilmann C, Yang JA, Hardy TA. Treatment with the glucagon receptor antagonist LY2409021 increases ambulatory blood pressure in patients with type 2 diabetes. Diabetes Obes Metab. 2017 Aug;19(8):1071-1077. doi: 10.1111/dom.12904. Epub 2017 Mar 27. PMID 28191913

RESULTS

PARTICIPANT FLOW:
Groups:
- LY2409021: 20 milligrams (mg) LY2409021 given orally once daily in the morning for 12 months (52 weeks). Participants remained on stable doses of metformin and sulfonylurea, as prescribed by their personal physician.
- Sitagliptin: 100 mg sitagliptin given orally once daily in the morning for 12 months (52 weeks). Participants remained on stable doses of metformin and sulfonylurea, as prescribed by their personal physician.
- Placebo: Placebo matching LY2409021 and sitagliptin given orally once daily in the morning for 12 months (52 weeks). Participants remained on stable doses of metformin and sulfonylurea, as prescribed by their personal physician.
Period: Overall Study
Arm/Group | LY2409021 | Sitagliptin | Placebo
Started | 65 | 41 | 68
Received at Least 1 Dose of Study Drug | 65 | 41 | 68
Completed | 1 | 0 | 2
Not Completed | 64 | 41 | 66
Not completed — Adverse Event | 4 | 1 | 2
Not completed — Non-Compliance with Study Drug | 1 | 1 | 0
Not completed — Lost to Follow Up | 1 | 1 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Terminated by Sponsor | 53 | 35 | 54
Not completed — Withdrawal by Subject | 4 | 2 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2409021 | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 65 | 41 | 68 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (8.33) | 57.1 (8.99) | 57.8 (8.21) | 57.3 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 10 | 31 | 65
  Male | 41 | 31 | 37 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 19 | 42 | 91
  Not Hispanic or Latino | 34 | 21 | 25 | 80
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 6 | 11 | 31
  White | 42 | 31 | 51 | 124
  More than one race | 5 | 2 | 1 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Greece | 6 | 4 | 6 | 16
  Puerto Rico | 8 | 5 | 13 | 26
  United States | 48 | 31 | 45 | 124
  Taiwan | 3 | 1 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 6 Months in Hepatic Fat Fraction
Description: The hepatic fat fraction (HFF) was calculated by a core imaging laboratory from noncontrast magnetic resonance imaging (MRI) of the liver. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, country, baseline HbA1c stratum (<=8.0%, >8.0%), visit, baseline score, and treatment-by-visit.
Time Frame: Baseline, 6 months
Population: All randomized participants who received at least 1 dose of study drug, have usable MRI HFF data at baseline and at least 1 post-baseline time point, excluding any data collected after stopping study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 62 | 39 | 67
percentage | 3.65 [2.13 to 5.17] | -0.07 [-1.94 to 1.79] | -0.79 [-2.28 to 0.70]

2. Secondary Outcome: Change From Baseline to 6 Months in Alanine Aminotransferase Levels
Description: Alanine aminotransferase (ALT) assessed by a central laboratory. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, country, baseline HbA1c stratum (<=8.0%, >8.0%), visit, baseline score, and treatment-by-visit.
Time Frame: Baseline, 6 months
Population: All randomized participants who received at least 1 dose of study drug, baseline data and at least 1 post-baseline time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: microgram per Liter (µ/L)
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 64 | 39 | 67
microgram per Liter (µ/L) | 9.4 [4.6 to 14.2] | 2.6 [-3.1 to 8.3] | -1.3 [-6.0 to 3.4]

3. Secondary Outcome: Number of Participants With Hepatobiliary Adverse Events of Special Interest (AESI)
Description: Number of participants with ALT or AST greater than 3 times the upper limit of normal at a post-baseline visit. A summary of other non-serious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Baseline, 6 months
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 65 | 41 | 68
Participants | 0 | 1 | 1

4. Secondary Outcome: Change From Baseline to 6 Months in Fasting Lipids Levels
Description: Lipid values (cholesterol, HDL cholesterol, LDL cholesterol, and triglycerides) assessed by a central laboratory. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, country, baseline HbA1c stratum (<=8.0%, >8.0%), visit, baseline score, and treatment-by-visit.
Time Frame: Baseline, 6 months
Population: All randomized participants who received at least 1 dose of randomized study drug, have data at baseline and at least 1 post-baseline time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimol per liter (mmol/L)
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 65 | 41 | 68
millimol per liter (mmol/L)
  Cholesterol: number analyzed (Participants) | 58 | 38 | 60
  Cholesterol | 0.468 [0.222 to 0.714] | 0.006 [-0.282 to 0.295] | 0.130 [-0.110 to 0.371]
  HDL Cholesterol: number analyzed (Participants) | 58 | 38 | 60
  HDL Cholesterol | 0.046 [-0.008 to 0.100] | 0.032 [-0.031 to 0.095] | -0.021 [-0.032 to 0.074]
  Triglycerides: number analyzed (Participants) | 58 | 38 | 60
  Triglycerides | 0.375 [0.087 to 0.644] | 0.078 [-0.264 to 0.420] | 0.099 [-0.183 to 0.381]
  LDL cholesterol: number analyzed (Participants) | 55 | 36 | 57
  LDL cholesterol | 0.244 [0.019 to 0.486] | -0.075 [-0.342 to 0.192] | 0.019 [-0.200 to 0.239]

5. Secondary Outcome: Change From Baseline to 6 Months in Fasting Blood Glucagon
Description: Glucagon values assessed by a central laboratory. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, country, baseline HbA1c stratum (<=8.0%, >8.0%), visit, baseline score, and treatment-by-visit.
Time Frame: Baseline, 6 months
Population: All randomized participants who received at least 1 dose of study drug, have data at baseline and at least 1 post-baseline time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: picomol per liter (pmol/L)
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 57 | 38 | 61
picomol per liter (pmol/L) | 44.06 [36.36 to 51.76] | 3.38 [-5.64 to 12.41] | 5.05 [-2.50 to 12.60]

6. Secondary Outcome: Change From Baseline to 6 Months in Body Weight
Description: Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, country, baseline HbA1c stratum (<=8.0%, >8.0%), visit, baseline score, and treatment-by-visit.
Time Frame: Baseline, 6 months
Population: as for outcome 5
Measure: Least Squares Mean (90% Confidence Interval); unit: kilograms (kg)
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 64 | 40 | 68
kilograms (kg) | 0.37 [0.12 to 0.63] | -0.08 [-0.39 to 0.22] | -0.05 [-0.30 to 0.20]

7. Secondary Outcome: Change From Baseline to 6 Months in Hemoglobin A1c (HbA1c)
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, country, visit, baseline score, and treatment-by-visit.
Time Frame: Baseline, 6 months
Population: All randomized participants who received at least 1 dose of study drug, have data at baseline and at least 1 post-baseline time point, excluding data collected after stopping study drug and/or starting rescue therapy.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent of HbA1c
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 63 | 40 | 68
percent of HbA1c | -0.63 [-0.94 to -0.32] | -0.42 [-0.80 to -0.05] | 0.14 [-0.15 to 0.45]

8. Secondary Outcome: Change From Baseline to 6 Months in Fasting Plasma Glucose
Description: as for outcome 6
Time Frame: Baseline, 6 months
Population: All randomized participants who received at least 1 dose of study drug,have data at baseline and at least 1 post-baseline time point, excluding data collected after stopping study drug and/or starting rescue therapy.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligram per decililiter (mg/dL)
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 63 | 40 | 61
milligram per decililiter (mg/dL) | -20.5 [-34.3 to -6.6] | -9.4 [-26.3 to 7.4] | 6.6 [-7.0 to 20.2]

9. Secondary Outcome: Change From Baseline to 6 Months in Blood Pressure
Description: Seated systolic blood pressure (SBP) and seated diastolic blood pressure (DBP) were measured in triplicate throughout the study. At each visit, all available blood pressure measurements for a subject were averaged to provide the blood pressure for that visit. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, country, baseline HbA1c stratum (<=8.0%, >8.0%), visit, baseline score, and treatment-by-visit.
Time Frame: Baseline, 6 months
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters of mercury (mm/Hg)
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 63 | 40 | 68
millimeters of mercury (mm/Hg)
  Systolic Blood Pressure | 6.1 [2.7 to 9.5] | 1.1 [-2.9 to 5.2] | 1.8 [-1.5 to 5.1]
  Diastolic Blood Pressure | 2.9 [0.7 to 5.0] | 0.3 [-2.3 to 2.9] | 1.5 [-0.6 to 3.6]

10. Secondary Outcome: Change From Baseline to 6 Months in Pulse Rate
Description: Seated pulse rate was measured in triplicate throughout the study. At each visit, all available pulse measurements for a subject were averaged to provide the pulse for that visit. Least Squares (LS) means were calculated using mixed model repeated measures (MMRM) adjusting for treatment, country, baseline HbA1c stratum (<=8.0%, >8.0%), visit, baseline score, and treatment-by-visit.
Time Frame: Baseline, 6 months
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: beats per minutes (bpm)
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 63 | 40 | 68
beats per minutes (bpm) | 1.5 [-0.6 to 3.7] | 3.5 [0.9 to 6.0] | 1.2 [-0.9 to 3.3]

11. Secondary Outcome: Change From Baseline to 6 Months in 7-Point Self-Monitoring of Blood Glucose (SMBG)
Description: 7-point profile consists of pre-meal and 2-hour postprandial SMBG measurements for the morning, midday, and evening meals in 1 day and at 3 AM (nocturnal blood glucose measurement). Pre-meal measurements were taken before the subject began eating the meal. Participants recorded their glucose measurements in their study diaries.
Time Frame: Baseline, 6 months
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 65 | 41 | 68
mg/dL
  Morning Pre-Meal: number analyzed (Participants) | 52 | 28 | 48
  Morning Pre-Meal | -29.4 (40.36) | -8.13 (31.25) | -4.31 (26.69)
  Mid-day Pre Meal: number analyzed (Participants) | 51 | 28 | 47
  Mid-day Pre Meal | -28.43 (41.13) | -30.58 (48.98) | -9.30 (51.08)
  Morning 2 Hour (Hr) Post Meal: number analyzed (Participants) | 48 | 28 | 44
  Morning 2 Hour (Hr) Post Meal | -38.8 (47.71) | -30.76 (44.35) | -18.28 (46.20)
  Midday 2 hr Post Meal: number analyzed (Participants) | 47 | 28 | 45
  Midday 2 hr Post Meal | -24.22 (52.64) | -25.20 (61.57) | -10.49 (54.17)
  Evening Pre Meal: number analyzed (Participants) | 51 | 28 | 47
  Evening Pre Meal | -24.58 (50.78) | -16.78 (51.09) | -14.13 (50.01)
  Evening 2 hr Post Meal: number analyzed (Participants) | 50 | 28 | 46
  Evening 2 hr Post Meal | -28.36 (58.92) | -21.12 (48.19) | -9.50 (48.62)
  Three AM: number analyzed (Participants) | 48 | 27 | 45
  Three AM | -22.78 (42.49) | -20.12 (57.39) | 0.88 (41.94)

12. Secondary Outcome: Population Pharmacokinetics: Apparent Clearance of LY2409021
Description: Reported as a Population Estimate with % Standard Errors of Estimation (SEE), 5th-95th confidence interval.
Time Frame: Day 1 Month 1, 3, 6, 9, predose, 1 hour postdose,
Population: All randomized participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Number (95% Confidence Interval); unit: Liters per hour (L/h)
Arm/Group | LY2409021
Number analyzed (Participants) | 65
Liters per hour (L/h) | 0.526 [0.454 to 0.598]

13. Secondary Outcome: Population Pharmacokinetics: Apparent Volume of Distribution of LY2409021
Time Frame: Day 1 Month 1, 3, 6, 9, predose, 1 hour postdose,
Population: All participants who received at least 1 dose of study drug and had evaluable PK data.
Measure: Number (95% Confidence Interval); unit: Liters (L)
Arm/Group | LY2409021
Number analyzed (Participants) | 65
Liters (L) | 31.9 [24.5 to 39.3]

14. Secondary Outcome: Rate of Hypoglycemic Events Adjusted Per 30 Days
Description: Documented symptomatic hypoglycemia, an event during which typical symptoms of hypoglycemia are accompanied by a measured plasma glucose concentration <=70 mg/dL (<=39 mmol/L),is presented. Rate: (30 days) is calculated as: (number of episodes during the time period divided by the number of days during the time period) multiplied by 30.
Time Frame: Baseline through 6 months
Population: as for outcome 7
Measure: Number; unit: number of episodes per day
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 64 | 40 | 68
number of episodes per day | 0.27 | 0.19 | 0.12

15. Secondary Outcome: Number of Participants With Hypoglycemic Events
Description: Documented symptomatic hypoglycemia, an event during which typical symptoms of hypoglycemia are accompanied by a measured plasma glucose concentration <=70 mg/dL (<=39 mmol/L), is presented. The number of subjects with an event are subjects who had at least one episode of documented symptomatic hypoglycemia during the time period.
Time Frame: Baseline through 6 months
Population: All randomized participants who received at least 1 dose of study drug, have data at baseline and at least 1 post-baseline time point, excluding data collected after study drug and/or starting rescue therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | LY2409021 | Sitagliptin | Placebo
Number analyzed (Participants) | 64 | 40 | 68
Participants | 20 | 40 | 68

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | LY2409021 | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 5/65 | 5/41 | 1/68
Other Adverse Events (participants affected / at risk) | 26/65 | 22/41 | 21/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2409021 (N=65) | Sitagliptin (N=41) | Placebo (N=68)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infectious colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2409021 (N=65) | Sitagliptin (N=41) | Placebo (N=68)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Type v hyperlipidaemia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 2 (2)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic retinal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Polyp (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Allergy to vaccine (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 2 (3) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (6) | 3 (3) | 3 (4)
Viral infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Free fatty acids increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Heart rate increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (5) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (8) | 2 (8) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Terminated, The overall benefit-risk profile did not support continued development of LY2409021 for type 2 diabetes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days